CLINICAL TRIAL: NCT01422031
Title: Utilization Pattern of Primary Health Care Services in Hong Kong - Does Having a Family Doctor Make Any Difference?
Brief Title: Study on Primary Care Health Service Utilization in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Cindy L.K. LAM, Head and Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-366
Record Dates: First submitted 2011-08-08; First posted 2011-08-23 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Primary Care; Health Services Utilization; Family Practice
Keywords: Primary care; Family doctor; Consultation; utilization; Non-drug managements; Patient enablement index
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Regular Family Doctor (RFD): People had a regular primary care doctor who is a family doctor
- Regular not Family doctor (RnFD): People had a regular primary care doctor who is not a family doctor
- Not regular doctor (NRD): People had no regular primary care doctor

SUMMARY:
The aim of this study was to find out the utilization rate and pattern of primary health care services, and the process and outcomes of primary care consultations of the general population in Hong Kong, and whether having a family doctor would make any difference.

The study objectives were to determine

1. the rates and pattern of utilization of different primary health care services and self-care
2. Patient self-reported outcomes (global rating on change in health, satisfaction and patient enablement) of primary care consultations;
3. the process of care in consultations including drug and non-drug managements, investigations, preventive care and referrals;
4. the effect of having a regular family doctor on service utilization rate and pattern, health promotion practice, and process and outcomes of primary care consultations.

DETAILED DESCRIPTION:
Study Design: A Cross-sectional general population survey and a longitudinal study (12-weeks follow up)

Method: Two phases, corresponding to Summer and Winter, respectively, of cross-sectional telephone survey on the Hong Kong general population using a structured questionnaire to collect information on the choice primary care doctors, illness rates, primary care service utilization rates and self-reported process and outcomes of consultations. A longitudinal study for 12 weeks was carried out on a sub-sample of the cross-sectional study subjects to collect data to cross-validate cross-sectional data. Univariate and multivariate regression analyses were used to determine whether there was any difference in service utilization rates, process and outcomes among people using different types of primary care doctors.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to study

Exclusion Criteria:

* Non-residential numbers
* Inability to communicate in Cantonese, Putonghua or English
* Refusal to telephone interview
* No contact after 5 attempts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 5174 eligible households were contacted by telephone but 1532 refused to be interviewed and 494 did not complete the interview. 3148 (60.8%) subjects, with 1616 and 1532 in the first and second phases, respectively, completed the cross-sectional survey. 1131 people (480 by additional telephone sampling) were invited to the longitudinal study but only 708 eventually agreed to take part and 327 returned the diaries (all by completion). 319 subjects had complete cross-sectional and longitudinal data for the final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 3148 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Primary care doctor choice group | baseline
Monthly utilization rate | Baseline
Patient Enablement Instrument (PEI) | Baseline
Rates of non-drug managements | Baseline

SECONDARY OUTCOMES:
Doctor shopping rate | Baseline
Self-medication rates during the last episode of illness | Baseline
Prescribing rate during last episode of illness | Baseline
Prevalence of preventive care | Baseline
Self-perceived health score | Baseline
Patient satisfaction | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Principal Investigator — Family Medicine Unit, Faculty of Medicine, HKU
Locations (1):
- Family Medicine Unit, Faculty of Medicine, HKU, Hong Kong, Hong Kong, China

REFERENCES:
- [Result] Lam CL, Leung GM, Mercer SW, Fong DY, Lee A, Lam TP, Lo YT. Utilisation patterns of primary health care services in Hong Kong: does having a family doctor make any difference? Hong Kong Med J. 2011 Jun;17(3 Suppl 3):28-32. No abstract available. PMID 21673357
- [Result] Lam CL, Yu EY, Lo YY, Wong CK, Mercer SM, Fong DY, Lee A, Lam TP, Leung GM. Having a Family Doctor is Associated with Some Better Patient-Reported Outcomes of Primary Care Consultations. Front Med (Lausanne). 2014 Sep 15;1:29. doi: 10.3389/fmed.2014.00029. eCollection 2014. PMID 25593904
- [Derived] Fung CS, Wong CK, Fong DY, Lee A, Lam CL. Having a family doctor was associated with lower utilization of hospital-based health services. BMC Health Serv Res. 2015 Jan 28;15:42. doi: 10.1186/s12913-015-0705-7. PMID 25627936